CLINICAL TRIAL: NCT06426069
Title: Assessment of Masticatory Performance in Various Stages of Periodontitis
Brief Title: Assessment of Masticatory Performance in Periodontitis
Status: Not yet recruiting | Type: Observational
Sponsor: Postgraduate Institute of Dental Sciences Rohtak (Other)
Responsible Party: Sponsor
Other Study IDs: JANVIPERIO2024
Record Dates: First submitted 2024-05-17; First posted 2024-05-23 (Actual); Last update posted 2024-05-23 (Actual); Status verified 2024-05

CONDITIONS: Periodontitis, Chronic; Chewing Problem; Inflammation
MeSH Terms: conditions — Chronic Periodontitis; Inflammation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (5):
- Periodontally Healthy: Complete periodontal examination will be done comprising of recording pocket probing depth (PPD), clinical attachment level (CAL) at six sites per tooth, bleeding on probing (BOP), plaque index (PI) and gingival index (GI) and mobility. Objective Masticatory Performance will be evaluated using colour mixing ability of a chewing gum. Subjective masticatory performance will be calculated using The Quality of Masticatory Function Questionnaire.
  Interventions: Other: Masticatory efficiency assessment
- Stage I Periodontitis: Complete periodontal examination will be done comprising of recording pocket probing depth (PPD), clinical attachment level (CAL) at six sites per tooth, bleeding on probing (BOP), plaque index (PI) and gingival index (GI) and mobility. Objective Masticatory Performance will be evaluated using colour mixing ability of a chewing gum. Subjective masticatory performance will be calculated using The Quality of Masticatory Function Questionnaire.
  Interventions: Other: Masticatory efficiency assessment
- Stage II Periodontitis: Complete periodontal examination will be done comprising of recording pocket probing depth (PPD), clinical attachment level (CAL) at six sites per tooth, bleeding on probing (BOP), plaque index (PI) and gingival index (GI) and mobility. Objective Masticatory Performance will be evaluated using colour mixing ability of a chewing gum. Subjective masticatory performance will be calculated using The Quality of Masticatory Function Questionnaire.
  Interventions: Other: Masticatory efficiency assessment
- Stage III Periodontitis: Complete periodontal examination will be done comprising of recording pocket probing depth (PPD), clinical attachment level (CAL) at six sites per tooth, bleeding on probing (BOP), plaque index (PI) and gingival index (GI) and mobility. Objective Masticatory Performance will be evaluated using colour mixing ability of a chewing gum. Subjective masticatory performance will be calculated using The Quality of Masticatory Function Questionnaire.
  Interventions: Other: Masticatory efficiency assessment
- Stage IV Periodontitis: Complete periodontal examination will be done comprising of recording pocket probing depth (PPD), clinical attachment level (CAL) at six sites per tooth, bleeding on probing (BOP), plaque index (PI) and gingival index (GI) and mobility. Objective Masticatory Performance will be evaluated using colour mixing ability of a chewing gum. Subjective masticatory performance will be calculated using The Quality of Masticatory Function Questionnaire.
  Interventions: Other: Masticatory efficiency assessment

INTERVENTIONS:
Other: Masticatory efficiency assessment — Masticatory efficiency will be assessed for each group.

SUMMARY:
The loss of periodontal attachment contributes to reduced masticatory performance and has a negative impact on general health.This clinical trial aims to assess the status of masticatory performance among patients with stage I, stage II, stage III and stage IV periodontitis, along with those with healthy periodontium.

DETAILED DESCRIPTION:
Periodontal disease manifestations include gingival bleeding, halitosis, tooth mobility and loss of teeth in advanced cases. The loss of periodontal attachment contributes to reduced masticatory performance and has a negative impact on general health. Loss of periodontium leads to reduced ability of tooth to withstand masticatory loads. Thus, biting abilities of subjects with healthy periodontium are significantly greater than those of chronic periodontitis patients. Even though the new periodontitis classification includes masticatory dysfunction in stage 4, but clinical periodontal parameters do start influencing objective masticatory efficiency in early stages. Since the masticatory function is an important point for the classification of periodontitis, standardized procedures with corresponding reference values are needed to consider these parameters in the assessment of periodontitis and to be able to make specific therapy recommendations.

This clinical trial aims to assess the changes in masticatory performance among periodontitis patients of all stages and healthy individuals using test methods easily applicable in daily practice.

ELIGIBILITY:
Inclusion Criteria:

1. Adult patients with age group 30-50 years diagnosed with generalized periodontitis
2. Presence of minimum 20 teeth (Eichner group A1, A2, A3) excluding third molars.

Exclusion Criteria:

* Systemic diseases that may affect periodontal disease progression or outcome of treatment (diabetes, autoimmune diseases)
* Systemic diseases that may affect masticatory ability of the patient (sarcopenia, TMJ disorders, Xerostomia, Acute Pulpitis)
* Grade C periodontitis (evaluated indirectly by radiographic bone loss/age criteria)
* Smoking or substance abuse
* Pregnant and lactating women

Ages: 30 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: A total of 555 patients will be recruited from the out patient department of periodontics, PGIDS, Rohtak based on the inclusion and exclusion criteria. The study design will be explained to eligible candidates and all study participants will be required to provide informed consent. Subjects will be grouped based on stage of periodontitis and a healthy control group.
Sampling Method: Probability Sample
Enrollment: 555 (Estimated)
Dates: Start 2024-06 (Estimated); Primary Completion 2024-12 (Estimated); Study Completion 2025-01 (Estimated)

PRIMARY OUTCOMES:
Objective masticatory performance | Baseline
  Objective Masticatory Performance will be evaluated using colour mixing ability of a chewing gum, through optoelectronic analysis using a software.

SECONDARY OUTCOMES:
Subjective masticatory performance | Baseline
  Subjective masticatory performance will be calculated using The Quality of Masticatory Function Questionnaire which consists of 29 questions related to frequency and difficulty of chewing different types of foods in the previous 2 weeks.

CONTACTS AND LOCATIONS:
Overall Officials: Janvi Janvi, BDS, Principal Investigator — PGIDS Rohtak
Locations (1):
- Post Graduate Institute of Dental Sciences, Rohtak, Haryana, India

IPD SHARING:
Plan to Share IPD: No